CLINICAL TRIAL: NCT03225287
Title: A Multicenter, Open-label, Uncontrolled, Extension Study of RA101495 in Subjects With Paroxysmal Nocturnal Hemoglobinuria Who Have Completed a RA101495 Clinical Study
Brief Title: Extension Study of RA101495 for Patients With PNH Who Have Completed a Zilucoplan (RA101495) Clinical Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After careful consideration, UCB has decided to no longer pursue PNH as a potential indication for zilucoplan.
Sponsor: Ra Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA101495-01.202; 2016-003523-34 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — zilucoplan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilucoplan (RA101495) (Experimental): Subjects will continue to receive the final maintenance dose they were receiving in the qualifying study
  Interventions: Drug: Zilucoplan (RA101495)

INTERVENTIONS:
Drug: Zilucoplan (RA101495) — Subjects will continue to receive the final maintenance dose they were receiving in the qualifying study.

SUMMARY:
The purpose of this study is to enable continued access to zilucoplan (RA101495) for patients with paroxysmal nocturnal hemoglobinuria (PNH) after they complete a zilucoplan clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a qualifying Ra Pharmaceuticals sponsored zilucoplan (RA101495) PNH study
* Evidence of ongoing clinical benefit in the opinion of the Investigator

Exclusion criteria:

* History of meningococcal disease
* Current systemic infection or suspicion of active bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anita Hill, Study Chair — St James' Institute of Oncology
Locations (12):
- United States (2):
  - Investigative Site 4, Los Angeles, California
  - Investigative Site 19, Dallas, Texas
- Australia (2):
  - Investigative Site 3, Gosford
  - Investigative Site 5, Melbourne
- Investigative Site 10, Toronto, Canada
- Investigative Site 14, Helsinki, Finland
- Investigative Site 9, Ulm, Germany
- Investigative Site 17, Budapest, Hungary
- New Zealand (2):
  - Investigative Site 13, Christchurch
  - Investigative Site 12, Hamilton
- United Kingdom (2):
  - Investigative Site 6, Leeds
  - Investigative Site 7, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Kulasekararaj AG, Lehtinen AE, Forsyth C, Gandhi S, Griffin M, Korper S, Mikala G, Muus P, Overgaard U, Patriquin CJ, Pullon H, Shen YM, Spearing R, Szer J, De la Borderie G, Duda PW, Farzaneh-Far R, Ragunathan S, Sayegh CE, Vadysirisack DD, Schrezenmeier H. Phase II trials of zilucoplan in paroxysmal nocturnal hemoglobinuria. Haematologica. 2024 Mar 1;109(3):929-935. doi: 10.3324/haematol.2022.281780. No abstract available. PMID 37534517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in July 2017 and concluded in October 2021.
Pre-assignment Details: The Participant Flow refers to the All Enrolled Subjects.
Groups:
- Zilucoplan-Cohort A (Eculizumab Naïve): Cohort A (Eculizumab Naive) included all participants from study RA101495-01.201 (NCT03078582) who had not received eculizumab for treatment of paroxysmal nocturnal hemoglobinuria (PNH). Participants received a loading dose of 0.3 milligram/kilogram (mg/kg) zilucoplan administered by subcutaneous (SC) injection at Day 1 of this study. Following in-clinic education and training, all participants self-injected 0.1 mg/kg of zilucoplan by SC injection once daily for 12 months. From Week 2 onwards, if a participant had not achieved an adequate response, the zilucoplan dose was escalated to 0.3 mg/kg daily.
- Zilucoplan-Cohort B (Eculizumab Switch): Cohort B (Eculizumab Switch) included all participants from study RA101495-01.201 (NCT03078582) who had received eculizumab for treatment of PNH. Participants received a loading dose of 0.3 mg/kg zilucoplan administered by SC injection at Day 1 of this study. Following in-clinic education and training, all participants self-injected 0.1 mg/kg of zilucoplan by SC injection once daily for 12 months. From Week 2 onwards, if a participant had not achieved an adequate response, the zilucoplan dose was escalated to 0.3 mg/kg daily.
- Zilucoplan (Inadequate Responder to Eculizumab): Inadequate Responder cohort included participants from qualifying study RA101495-01.203 (NCT03030183) who had an inadequate response to eculizumab treatment for PNH. Participants received a loading dose of 0.3 mg/kg zilucoplan administered by SC injection at Day 1 of this study. Following in-clinic education and training, all participants self-injected 0.1 mg/kg of zilucoplan by SC injection once daily for 12 months. From Week 2 onwards, if a participant had not achieved an adequate response, the zilucoplan dose was escalated to 0.3 mg/kg daily.
Period: Overall Study
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Started | 10 | 6 | 3
Completed | 0 | 0 | 0
Not Completed | 10 | 6 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol non-compliance | 0 | 0 | 1
Not completed — Subject withdraws consent | 3 | 0 | 0
Not completed — Sponsor, regulatory, or EC/IRB request | 7 | 3 | 1
Not completed — Trial drug not effective | 0 | 1 | 0
Not completed — Need of transfusions and signs of hemolysis | 0 | 1 | 0
Not completed — Stem cell transplantation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Population which consisted of all participants who received at least 1 injection of zilucoplan on or after Day 1 of the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab) | Total
Number analyzed (Participants) | 10 | 6 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 3 | 13
  >=65 years | 4 | 2 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (14.5) | 45.0 (23.0) | 35.3 (16.3) | 51.2 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 1 | 8
  Male | 4 | 5 | 2 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 6 | 1 | 17
  Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 10 | 5 | 3 | 18
  Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as an AE that occurs after a participant's initial treatment zilucoplan start for this study (RA101495-01.202) that was not present at the time of treatment start, or an AE that increases in severity after treatment start in this study, if the event was present at the time of treatment start.
Time Frame: From Day 1 until the Final Study Visit (up to Month 49)
Population: Safety population included all participants who received at least 1 injection of zilucoplan on or after Day 1 of this extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 10 | 6 | 3
percentage of participants | 90.0 | 100 | 66.7

2. Primary Outcome: Percentage of Participants With Serious TEAEs
Description: Serious Adverse event (SAE) was defined as any untoward medical occurrence that:• results in death, • is life-threatening threatening (note that this refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe), • requires hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity, and • results in a congenital anomaly/birth defect.
Time Frame: From Day 1 until the Final Study Visit (up to Month 49)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 10 | 6 | 3
percentage of participants | 10.0 | 50.0 | 66.7

3. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: Blood samples collection were planned to analyze for the presence/absence of ADAs to zilucoplan for immunogenicity assessments.
Time Frame: At Day 1, Month 1, 2, 3, 6, 9, and 12
Population: Safety population included all participants who received at least 1 injection of zilucoplan on or after Day 1 of this extension study. The planned analysis of immunogenicity (ADA) was not performed as the assay was considered not fit for purpose due to an insufficient level of drug tolerance; therefore, no samples were processed.
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Serum Lactate Dehydrogenase (LDH) Levels at Each Time Point
Description: Serum LDH levels were measure of intravascular hemolysis. As high level of LDH in the blood was indicative of hemolysis in participants with PNH.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: Safety population included all participants who received at least 1 injection of zilucoplan on or after Day 1 of this extension study. Baseline was generally the final visit of the qualifying study (RA101495-01.201 or RA101495-01.203). Here, Number of participants analyzed included those participants who were evaluable for the assessment and 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
Units per litre (U/L)
  Month 1 | -3.7 (71.5) | 10.0 (16.4) | 336.7 (636.9)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 50.3 (156.2) | -2.4 (22.2) | 676.5 (970.9)
  Month 3: number analyzed (Participants) | 8 | 5 | 2
  Month 3 | -6.5 (58.2) | -1.6 (40.5) | 39.5 (40.3)
  Month 6: number analyzed (Participants) | 8 | 5 | 2
  Month 6 | 32.4 (142.5) | -28.4 (127.3) | -3.5 (12.0)
  Month 9: number analyzed (Participants) | 8 | 3 | 2
  Month 9 | -18.1 (59.7) | 22.7 (23.6) | -5.0 (35.4)
  Month 12: number analyzed (Participants) | 7 | 3 | 2
  Month 12 | -39.7 (54.9) | 8.7 (10.1) | 456.0 (640.6)
  Month 15: number analyzed (Participants) | 6 | 3 | 2
  Month 15 | -24.5 (70.8) | 4.0 (30.4) | 174.5 (215.7)
  Month 18: number analyzed (Participants) | 7 | 3 | 1
  Month 18 | -27.9 (54.8) | 5.7 (56.8) | -56.0 (NA) — Standard Deviation (SD) could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 1
  Month 21 | -12.0 (93.9) | -7.3 (33.5) | 73.0 (NA) — SD could not be calculated for a single participant.
  Month 24: number analyzed (Participants) | 7 | 3 | 1
  Month 24 | -18.7 (53.9) | -27.0 (64.1) | -29.0 (NA) — SD could not be calculated for a single participant.
  Month 27: number analyzed (Participants) | 5 | 2 | 0
  Month 27 | -14.0 (99.3) | 58.0 (8.5) |
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | -28.0 (36.1) | 59.0 (140.0) | 1817.0 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | -39.0 (65.9) | -16.3 (66.7) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | -61.6 (47.1) | 0.5 (4.9) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | -78.4 (80.9) | -29.7 (83.5) |
  Month 42: number analyzed (Participants) | 4 | 2 | 0
  Month 42 | -42.3 (78.3) | 35.5 (75.7) |
  Month 45: number analyzed (Participants) | 1 | 1 | 0
  Month 45 | 27.0 (NA) — SD could not be calculated for a single participant. | 53.0 (NA) — SD could not be calculated for a single participant. |
  Final Study Visit (Month 49): number analyzed (Participants) | 9 | 5 | 2
  Final Study Visit (Month 49) | 41.6 (303.1) | -93.2 (139.8) | 682.0 (548.7)

5. Secondary Outcome: Change From Baseline in Total Bilirubin Values at Each Time Point
Description: Total Bilirubin was monitored for signs and symptoms of hepatic or biliary dysfunction.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromole per litre (umol/L)
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
micromole per litre (umol/L)
  Month 1 | -2.1 (7.7) | 1.7 (6.2) | -0.3 (4.5)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 0.1 (10.7) | 2.0 (7.2) | 6.0 (2.8)
  Month 3: number analyzed (Participants) | 8 | 5 | 2
  Month 3 | 1.4 (13.7) | 8.2 (13.1) | 3.5 (2.1)
  Month 6: number analyzed (Participants) | 8 | 5 | 2
  Month 6 | 4.6 (14.8) | 3.2 (7.2) | 2.5 (0.7)
  Month 9: number analyzed (Participants) | 8 | 3 | 2
  Month 9 | -0.3 (7.4) | 6.0 (3.0) | -1.0 (1.4)
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | 3.9 (8.4) | 3.0 (2.0) | 2.5 (3.5)
  Month 15: number analyzed (Participants) | 7 | 3 | 2
  Month 15 | -0.4 (6.4) | 6.0 (9.5) | 8.5 (9.2)
  Month 18: number analyzed (Participants) | 6 | 3 | 1
  Month 18 | 2.8 (9.5) | 2.0 (6.2) | 3.0 (NA) — SD could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 1
  Month 21 | 3.9 (8.3) | 2.0 (7.8) | 7.0 (NA) — SD could not be calculated for a single participant.
  Month 24: number analyzed (Participants) | 7 | 3 | 1
  Month 24 | 5.1 (16.0) | -1.3 (3.1) | 8.0 (NA) — SD could not be calculated for a single participant.
  Month 27: number analyzed (Participants) | 7 | 2 | 0
  Month 27 | 4.3 (12.2) | -2.0 (5.7) |
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | 5.8 (14.6) | 3.0 (7.1) | 13.0 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | 2.6 (5.7) | 3.0 (2.6) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | -3.8 (6.8) | 3.0 (0.0) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | 0.2 (3.1) | 0.7 (4.6) |
  Month 42: number analyzed (Participants) | 5 | 2 | 0
  Month 42 | 4.8 (15.5) | 4.0 (15.6) |
  Month 45: number analyzed (Participants) | 2 | 1 | 0
  Month 45 | 5.0 (17.0) | -2.0 (NA) — SD could not be calculated for a single participant. |
  Final Study Visit (Month 49): number analyzed (Participants) | 9 | 5 | 2
  Final Study Visit (Month 49) | 8.0 (17.3) | 0.4 (3.9) | 0.0 (9.9)

6. Secondary Outcome: Change From Baseline in Total Hemoglobin Values at Each Time Point
Description: Total Hemoglobin Values were analyzed for hematology assessments.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
grams per litre (g/L)
  Month 1: number analyzed (Participants) | 8 | 6 | 3
  Month 1 | 0.0 (11.4) | 0.0 (8.2) | -5.7 (3.8)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 1.1 (8.3) | -5.0 (9.9) | -2.0 (11.3)
  Month 3: number analyzed (Participants) | 7 | 5 | 2
  Month 3 | 6.4 (6.4) | 3.0 (9.1) | -3.5 (6.4)
  Month 6: number analyzed (Participants) | 8 | 5 | 2
  Month 6 | 1.1 (11.2) | 2.0 (17.9) | -5.0 (17.0)
  Month 9: number analyzed (Participants) | 8 | 3 | 2
  Month 9 | 2.9 (7.1) | -1.3 (4.0) | -9.0 (5.7)
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | 2.9 (6.1) | -1.7 (6.8) | -5.0 (17.0)
  Month 15: number analyzed (Participants) | 7 | 3 | 2
  Month 15 | 3.9 (8.4) | -5.0 (5.3) | -9.0 (28.3)
  Month 18: number analyzed (Participants) | 7 | 3 | 1
  Month 18 | 5.0 (4.9) | 1.7 (9.5) | -2.0 (NA) — SD could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 1
  Month 21 | 6.4 (6.3) | -6.7 (7.6) | -1.0 (NA) — SD could not be calculated for a single participant.
  Month 24: number analyzed (Participants) | 7 | 3 | 0
  Month 24 | 7.9 (12.6) | -5.0 (2.6) |
  Month 27: number analyzed (Participants) | 7 | 2 | 0
  Month 27 | 7.0 (10.0) | -5.0 (11.3) |
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | 10.8 (7.0) | -4.5 (12.0) | -8.0 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | 10.0 (8.8) | -3.0 (4.4) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | 8.4 (14.2) | -2.0 (4.2) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | 7.6 (10.1) | 4.7 (2.9) |
  Month 42: number analyzed (Participants) | 5 | 2 | 0
  Month 42 | 5.2 (11.2) | 5.5 (0.7) |
  Month 45: number analyzed (Participants) | 3 | 1 | 0
  Month 45 | -1.3 (23.3) | -4.0 (NA) — SD could not be calculated for a single participant. |
  Final Study Visit (Month 49): number analyzed (Participants) | 9 | 4 | 1
  Final Study Visit (Month 49) | 1.8 (10.6) | -2.0 (4.1) | -7.0 (NA) — SD could not be calculated for a single participant.

7. Secondary Outcome: Change From Baseline in Free Hemoglobin Values at Each Time Point
Description: Free Hemoglobin Values were analyzed for hematology assessments.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 7 | 5 | 2
milligrams per decilitre (mg/dL)
  Month 1: number analyzed (Participants) | 6 | 5 | 2
  Month 1 | -0.20 (2.78) | 2.86 (4.30) | 0.80 (4.38)
  Month 2: number analyzed (Participants) | 5 | 5 | 1
  Month 2 | -1.14 (3.04) | 0.48 (1.77) | 6.10 (NA) — SD could not be calculated for a single participant.
  Month 3: number analyzed (Participants) | 5 | 5 | 1
  Month 3 | 1.34 (0.48) | -0.02 (0.95) | 0.80 (NA) — SD could not be calculated for a single participant.
  Month 6: number analyzed (Participants) | 6 | 4 | 1
  Month 6 | -0.43 (1.24) | 0.55 (2.45) | 1.20 (NA) — SD could not be calculated for a single participant.
  Month 9: number analyzed (Participants) | 6 | 3 | 1
  Month 9 | -1.10 (2.11) | -1.50 (1.57) | 0.00 (NA) — SD could not be calculated for a single participant.
  Month 12: number analyzed (Participants) | 7 | 2 | 1
  Month 12 | -0.56 (2.80) | 0.80 (0.28) | 2.10 (NA) — SD could not be calculated for a single participant.
  Month 15: number analyzed (Participants) | 4 | 2 | 1
  Month 15 | 3.93 (11.61) | -1.35 (2.19) | 1.60 (NA) — SD could not be calculated for a single participant.
  Month 18: number analyzed (Participants) | 4 | 3 | 0
  Month 18 | 1.98 (3.05) | 0.77 (1.56) |
  Month 21: number analyzed (Participants) | 4 | 2 | 0
  Month 21 | 3.15 (5.84) | -1.30 (0.85) |
  Month 24: number analyzed (Participants) | 3 | 2 | 0
  Month 24 | 0.27 (0.35) | -0.50 (0.99) |
  Month 27: number analyzed (Participants) | 0 | 0 | 0
  Month 30: number analyzed (Participants) | 3 | 0 | 0
  Month 30 | 0.33 (2.37) |  |
  Month 33: number analyzed (Participants) | 3 | 1 | 0
  Month 33 | 0.17 (2.66) | 5.80 (NA) — SD could not be calculated for a single participant. |
  Month 36: number analyzed (Participants) | 0 | 0 | 0
  Month 39: number analyzed (Participants) | 1 | 2 | 0
  Month 39 | -0.60 (NA) — SD could not be calculated for a single participant. | -0.95 (0.64) |
  Month 42: number analyzed (Participants) | 1 | 2 | 0
  Month 42 | 1.30 (NA) — SD could not be calculated for a single participant. | 0.50 (3.68) |
  Month 45: number analyzed (Participants) | 0 | 0 | 0
  Final Study Visit (Month 49): number analyzed (Participants) | 1 | 2 | 1
  Final Study Visit (Month 49) | -2.70 (NA) — SD could not be calculated for a single participant. | -0.60 (1.13) | -3.10 (NA) — SD could not be calculated for a single participant.

8. Secondary Outcome: Change From Baseline in Haptoglobin Values at Each Time Point
Description: Haptoglobin values were analyzed for hematology assessments.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
g/L
  Month 1 | 0.032 (0.097) | 0.000 (0.000) | 0.000 (0.000)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 0.053 (0.160) | 0.000 (0.000) | 0.000 (0.000)
  Month 3: number analyzed (Participants) | 8 | 5 | 2
  Month 3 | 0.021 (0.060) | 0.000 (0.000) | 0.000 (0.000)
  Month 6: number analyzed (Participants) | 8 | 5 | 2
  Month 6 | 0.031 (0.088) | 0.036 (0.080) | 0.020 (0.028)
  Month 9: number analyzed (Participants) | 8 | 3 | 2
  Month 9 | 0.008 (0.021) | 0.000 (0.000) | 0.000 (0.000)
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Month 15: number analyzed (Participants) | 7 | 3 | 2
  Month 15 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Month 18: number analyzed (Participants) | 7 | 3 | 1
  Month 18 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (NA) — SD could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 1
  Month 21 | 0.030 (0.079) | 0.000 (0.000) | 0.000 (NA) — SD could not be calculated for a single participant.
  Month 24: number analyzed (Participants) | 7 | 3 | 1
  Month 24 | 0.030 (0.079) | 0.000 (0.000) | 0.000 (NA) — SD could not be calculated for a single participant.
  Month 27: number analyzed (Participants) | 7 | 2 | 0
  Month 27 | 0.000 (0.000) | 0.000 (0.000) |
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | 0.004 (0.009) | 0.000 (0.000) | 0.000 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | 0.002 (0.004) | 0.000 (0.000) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | 0.036 (0.080) | 0.000 (0.000) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | 0.020 (0.045) | 0.000 (0.000) |
  Month 42: number analyzed (Participants) | 5 | 2 | 0
  Month 42 | 0.034 (0.076) | 0.000 (0.000) |
  Month 45: number analyzed (Participants) | 2 | 1 | 0
  Month 45 | 0.080 (0.113) | 0.000 (NA) — SD could not be calculated for a single participant. |
  Final Study Visit (Month 49): number analyzed (Participants) | 9 | 5 | 2
  Final Study Visit (Month 49) | 0.042 (0.127) | 0.006 (0.013) | 0.000 (0.000)

9. Secondary Outcome: Change From Baseline in Reticulocytes at Each Time Point
Description: Reticulocytes values were analyzed for hematology assessments.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and Final Study Visit (Month 49)
Population: Safety population included all participants who received at least 1 injection of zilucoplan on or after Day 1 of this extension study. Here, Number of participants analyzed included those participants who were evaluable for the assessment and 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: 10^12 reticulocytes (cells)/L
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
10^12 reticulocytes (cells)/L
  Month 1: number analyzed (Participants) | 8 | 6 | 3
  Month 1 | 0.0104 (0.0484) | 0.0107 (0.0299) | -0.0457 (0.0505)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | -0.0046 (0.0354) | -0.0046 (0.0130) | 0.0115 (0.0049)
  Month 3: number analyzed (Participants) | 7 | 5 | 2
  Month 3 | -0.0249 (0.0310) | -0.0112 (0.0251) | 0.0170 (0.0113)
  Month 6: number analyzed (Participants) | 8 | 5 | 2
  Month 6 | -0.0006 (0.0452) | -0.0042 (0.0363) | 0.0200 (0.0382)
  Month 9: number analyzed (Participants) | 8 | 3 | 2
  Month 9 | 0.0063 (0.0334) | 0.0070 (0.0171) | 0.0640 (0.0297)
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | -0.0041 (0.0427) | -0.0070 (0.0346) | 0.0240 (0.0113)
  Month 15: number analyzed (Participants) | 7 | 3 | 2
  Month 15 | -0.0264 (0.0601) | -0.0343 (0.0191) | 0.0285 (0.0290)
  Month 18: number analyzed (Participants) | 7 | 3 | 1
  Month 18 | -0.0040 (0.0382) | 0.0027 (0.0380) | 0.0460 (NA) — SD could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 0
  Month 21 | -0.0223 (0.0554) | -0.0087 (0.0380) |
  Month 24: number analyzed (Participants) | 7 | 3 | 0
  Month 24 | -0.0123 (0.0711) | -0.0093 (0.0186) |
  Month 27: number analyzed (Participants) | 7 | 2 | 0
  Month 27 | -0.0017 (0.0553) | 0.0150 (0.0127) |
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | 0.0016 (0.0524) | 0.0060 (0.0594) | 0.0300 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | -0.0302 (0.0446) | -0.0093 (0.0234) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | -0.0630 (0.0621) | -0.0215 (0.0078) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | -0.0340 (0.0860) | -0.0133 (0.0291) |
  Month 42: number analyzed (Participants) | 5 | 2 | 0
  Month 42 | -0.0270 (0.0721) | -0.0015 (0.0078) |
  Month 45: number analyzed (Participants) | 3 | 1 | 0
  Month 45 | -0.0423 (0.1189) | -0.0050 (NA) — SD could not be calculated for a single participant. |
  Final Study Visit (Month 49): number analyzed (Participants) | 8 | 4 | 1
  Final Study Visit (Month 49) | -0.0433 (0.0480) | -0.0333 (0.0116) | 0.0100 (NA) — SD could not be calculated for a single participant.

10. Secondary Outcome: Change From Baseline in Hemoglobinuria Values at Each Time Point
Description: Hemoglobinuria was assessed using a urine colorimetric scoring system with a score of 1 through 10 where 1 represents no hemoglobinuria and 10 represents maximum hemoglobinuria.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48 and Final Study Visit (Month 49)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
score on a scale
  Month 1: number analyzed (Participants) | 8 | 6 | 3
  Month 1 | 0.1 (1.0) | 0.2 (1.5) | 1.7 (1.5)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 0.9 (1.4) | 0.8 (1.3) | 1.0 (1.4)
  Month 3: number analyzed (Participants) | 8 | 5 | 1
  Month 3 | 0.4 (1.2) | 0.8 (1.3) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 6: number analyzed (Participants) | 8 | 5 | 1
  Month 6 | 0.4 (0.9) | 0.8 (1.3) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 9: number analyzed (Participants) | 8 | 2 | 1
  Month 9 | 0.4 (0.9) | 1.5 (2.1) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | 0.9 (1.4) | 1.0 (1.7) | 1.0 (1.4)
  Month 15: number analyzed (Participants) | 7 | 3 | 2
  Month 15 | 0.9 (1.1) | 1.0 (1.7) | 1.0 (1.4)
  Month 18: number analyzed (Participants) | 7 | 3 | 1
  Month 18 | 0.1 (0.9) | 0.3 (0.6) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 21: number analyzed (Participants) | 7 | 3 | 1
  Month 21 | 0.7 (1.6) | 1.0 (1.7) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 24: number analyzed (Participants) | 7 | 3 | 1
  Month 24 | 0.6 (1.6) | 0.3 (0.6) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 27: number analyzed (Participants) | 7 | 2 | 1
  Month 27 | 0.7 (1.5) | 1.5 (2.1) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 30: number analyzed (Participants) | 5 | 2 | 1
  Month 30 | 0.6 (1.3) | 1.5 (2.1) | 0.0 (NA) — SD could not be calculated for a single participant.
  Month 33: number analyzed (Participants) | 5 | 3 | 0
  Month 33 | 1.4 (0.9) | 1.0 (1.7) |
  Month 36: number analyzed (Participants) | 5 | 2 | 0
  Month 36 | 1.4 (1.9) | 1.5 (2.1) |
  Month 39: number analyzed (Participants) | 5 | 3 | 0
  Month 39 | 0.4 (1.7) | 1.0 (1.7) |
  Month 42: number analyzed (Participants) | 5 | 2 | 0
  Month 42 | 1.0 (1.2) | 1.5 (2.1) |
  Month 45: number analyzed (Participants) | 3 | 1 | 0
  Month 45 | 1.0 (1.0) | -1.0 (NA) — SD could not be calculated for a single participant. |
  Month 48: number analyzed (Participants) | 0 | 0 | 0
  Final Study Visit (Month 49): number analyzed (Participants) | 9 | 5 | 2
  Final Study Visit (Month 49) | 0.4 (1.1) | 0.6 (0.9) | 2.5 (3.5)

11. Secondary Outcome: Plasma Concentrations of RA101495 and Its Major Metabolite(s)
Description: Blood samples of RA101495 (zilucoplan) and its metabolites (RA102758 and RA103488) were collected for Plasma concentration analysis.
Time Frame: Predose: At Day 1 (Screening), Month 1, 2, 3, 6, 9, 12, and Final Study Visit (Month 49)
Population: Pharmacokinetic (PK) population included all participants in the Safety population who had at least 1 plasma sample obtained for PK assessment. Here, 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: micrograms per litre (ug/L)
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 3
micrograms per litre (ug/L)
  RA101495- Day 1: number analyzed (Participants) | 9 | 5 | 3
  RA101495- Day 1 | 10999.99 (2698.29) | 13616.08 (1490.81) | 6976.50 (5663.23)
  RA101495- Month 1 | 10879.13 (2405.19) | 12645.38 (1620.31) | 7630.03 (7060.56)
  RA101495- Month 2: number analyzed (Participants) | 9 | 5 | 2
  RA101495- Month 2 | 11276.17 (2896.98) | 12220.10 (2188.78) | 6865.45 (8108.18)
  RA101495- Month 3: number analyzed (Participants) | 8 | 5 | 2
  RA101495- Month 3 | 10806.17 (3418.92) | 12315.28 (2515.84) | 12430.00 (16.55)
  RA101495- Month 6: number analyzed (Participants) | 6 | 5 | 1
  RA101495- Month 6 | 9393.42 (2224.52) | 12218.72 (2166.05) | 12254.00 (NA) — SD could not be calculated for a single participant.
  RA101495- Month 9: number analyzed (Participants) | 7 | 3 | 2
  RA101495- Month 9 | 11848.67 (2685.92) | 12282.83 (3064.42) | 15193.35 (2756.66)
  RA101495- Month 12: number analyzed (Participants) | 8 | 3 | 2
  RA101495- Month 12 | 11495.99 (2885.81) | 13279.97 (2148.60) | 12038.65 (7934.94)
  RA101495- Final Study Visit (Month 49): number analyzed (Participants) | 0 | 0 | 1
  RA101495- Final Study Visit (Month 49) |  |  | 7174.20 (NA) — SD could not be calculated for a single participant.
  RA102758- Day 1: number analyzed (Participants) | 9 | 5 | 3
  RA102758- Day 1 | 1883.49 (593.93) | 2443.62 (560.97) | 1280.07 (1109.03)
  RA102758- Month 1 | 1865.06 (594.31) | 2185.00 (631.37) | 757.30 (997.44)
  RA102758- Month 2: number analyzed (Participants) | 9 | 5 | 2
  RA102758- Month 2 | 1894.86 (608.46) | 2090.04 (831.80) | 757.85 (1018.59)
  RA102758- Month 3: number analyzed (Participants) | 8 | 5 | 2
  RA102758- Month 3 | 1758.55 (689.03) | 1990.54 (700.70) | 1954.05 (160.58)
  RA102758- Month 6: number analyzed (Participants) | 6 | 5 | 1
  RA102758- Month 6 | 1467.85 (563.68) | 1819.20 (613.14) | 1725.50 (NA) — SD could not be calculated for a single participant.
  RA102758- Month 9: number analyzed (Participants) | 7 | 3 | 2
  RA102758- Month 9 | 1686.80 (554.87) | 1881.73 (583.87) | 1238.55 (166.24)
  RA102758- Month 12: number analyzed (Participants) | 8 | 3 | 1
  RA102758- Month 12 | 1646.99 (536.00) | 1954.23 (725.54) | 10.00 (NA) — SD could not be calculated for a single participant.
  RA102758- Final Study Visit (Month 49): number analyzed (Participants) | 0 | 0 | 1
  RA102758- Final Study Visit (Month 49) |  |  | 1094.60 (NA) — SD could not be calculated for a single participant.
  RA103488- Day 1: number analyzed (Participants) | 9 | 5 | 3
  RA103488- Day 1 | 3587.68 (1747.12) | 4887.98 (1969.22) | 2084.83 (1791.35)
  RA103488- Month 1 | 4344.99 (2319.10) | 4400.68 (1823.93) | 1703.73 (1605.96)
  RA103488- Month 2: number analyzed (Participants) | 9 | 5 | 2
  RA103488- Month 2 | 4799.29 (3113.57) | 4365.84 (1537.67) | 1591.35 (1552.03)
  RA103488- Month 3: number analyzed (Participants) | 8 | 5 | 2
  RA103488- Month 3 | 4191.36 (2347.65) | 4541.78 (1706.07) | 2715.60 (1345.48)
  RA103488- Month 6: number analyzed (Participants) | 6 | 5 | 1
  RA103488- Month 6 | 4027.53 (2730.92) | 4436.46 (2341.16) | 1929.60 (NA) — SD could not be calculated for a single participant.
  RA103488- Month 9: number analyzed (Participants) | 7 | 3 | 2
  RA103488- Month 9 | 3132.54 (1320.61) | 4217.97 (2015.36) | 2954.85 (1754.97)
  RA103488- Month 12: number analyzed (Participants) | 8 | 3 | 2
  RA103488- Month 12 | 3903.41 (1960.30) | 4334.47 (1976.47) | 2319.20 (2534.84)
  RA103488- Final Study Visit (Month 49): number analyzed (Participants) | 0 | 0 | 1
  RA103488- Final Study Visit (Month 49) |  |  | 2210.00 (NA) — SD could not be calculated for a single participant.

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of RA101495
Description: Cmax is the maximum plasma concentration.
Time Frame: At Day 1, Month 1, 2, 3, 6, 9, and 12
Population: PK population included all participants in the Safety population who had at least 1 plasma sample obtained for PK assessment. Data was not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Time Corresponding to Cmax (Tmax) of RA101495
Description: tmax is the time to corresponding Cmax.
Time Frame: At Day 1, Month 1, 2, 3, 6, 9, and 12
Population: as for outcome 12
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Area Under the Drug Concentration-time Curve (AUC0-t) of RA101495
Description: AUC0-t is area under the drug concentration-time curves.
Time Frame: At Day 1, Month 1, 2, 3, 6, 9, and 12
Population: PK population included all participants in the Safety population who had at least 1 plasma sample obtained for PK assessment. As per the change in planned analyses, samples/data were not collected, and AUC0-t not calculated.
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Total Complement (CH50) Levels
Description: Blood samples collection were planned to assess complement (CH50) levels. The planned analysis of CH50 was not performed because the CH50 assay was not able to be validated due to lack of reproducibility of the manufacturer's kits.
Time Frame: At Day 1, Month 1, 2, 3, 6, 9, and 12
Population: Pharmacodynamic (PD) population included all participants in the Safety population who had at least 1 plasma sample obtained for PD assessment. Data was not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Sheep Red Blood Cell (sRBC) Values at Each Time Point
Description: Blood samples were collected for measurement of sRBC lysis for the Classical Complement Pathways.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12 and Final Study Visit (Month 49)
Population: PD population included all participants in the Safety population who had at least 1 plasma sample obtained for PD assessment. Here, Number of participants analyzed included those participants who were evaluable for the assessment and 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent lysis of sheep erythrocytes
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 1
percent lysis of sheep erythrocytes
  Month 1 | 1.378 (2.277) | 0.523 (0.772) | 93.870 (NA) — SD could not be calculated for a single participant.
  Month 2: number analyzed (Participants) | 9 | 5 | 1
  Month 2 | 1.248 (1.789) | -0.308 (0.452) | 93.870 (NA) — SD could not be calculated for a single participant.
  Month 3: number analyzed (Participants) | 8 | 5 | 1
  Month 3 | 1.256 (1.799) | 0.576 (0.972) | -2.620 (NA) — SD could not be calculated for a single participant.
  Month 6: number analyzed (Participants) | 6 | 5 | 1
  Month 6 | 1.493 (2.838) | 0.458 (1.657) | -2.300 (NA) — SD could not be calculated for a single participant.
  Month 9: number analyzed (Participants) | 7 | 3 | 1
  Month 9 | 0.683 (1.055) | 0.757 (0.673) | -1.410 (NA) — SD could not be calculated for a single participant.
  Month 12: number analyzed (Participants) | 8 | 3 | 1
  Month 12 | 0.759 (0.557) | 0.773 (0.415) | 8.390 (NA) — SD could not be calculated for a single participant.
  Final Study Visit (Month 49): number analyzed (Participants) | 0 | 2 | 0
  Final Study Visit (Month 49) |  | 25.230 (35.200) |

17. Secondary Outcome: Change From Baseline in Wieslab Enzyme-linked Immunosorbent Assay (ELISA) Values for Alternative Complement Pathway at Each Time Point
Description: Blood samples were collected for measurement of membrane attack complex (MAC) by Wieslab ELISA for alternative complement pathway.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12 and Final Study Visit (Month 49)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 2
percentage of activity
  Month 1 | 1.7 (5.8) | 1.0 (1.7) | 48.0 (67.9)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | 0.1 (1.9) | -1.0 (1.0) | 51.5 (74.2)
  Month 3: number analyzed (Participants) | 8 | 5 | 2
  Month 3 | 0.1 (2.0) | 0.0 (0.7) | 2.0 (1.4)
  Month 6: number analyzed (Participants) | 6 | 5 | 1
  Month 6 | 1.0 (4.5) | -0.2 (1.9) | 5.0 (NA) — SD could not be calculated for a single participant.
  Month 9: number analyzed (Participants) | 8 | 3 | 1
  Month 9 | -0.9 (0.8) | -0.7 (0.6) | -2.0 (NA) — SD could not be calculated for a single participant.
  Month 12: number analyzed (Participants) | 8 | 3 | 2
  Month 12 | -1.4 (1.4) | -1.3 (0.6) | 4.5 (6.4)
  Final Study Visit (Month 49): number analyzed (Participants) | 0 | 2 | 0
  Final Study Visit (Month 49) |  | 1.0 (2.8) |

18. Secondary Outcome: Change From Baseline in Complement Component 5 (C5) Values at Each Time Point
Description: Blood samples were collected for measurement of Complement component 5 (C5) levels.
Time Frame: Baseline, Month 1, 2, 3, 6, 9, 12 and Final Study Visit (Month 49)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
Number analyzed (Participants) | 9 | 6 | 2
ug/mL
  Month 1 | -11.231 (24.960) | 20.488 (31.024) | -27.505 (90.092)
  Month 2: number analyzed (Participants) | 9 | 5 | 2
  Month 2 | -15.914 (32.737) | 17.716 (33.125) | 16.310 (36.077)
  Month 3: number analyzed (Participants) | 8 | 5 | 2
  Month 3 | -24.404 (50.084) | -2.898 (49.747) | 22.355 (19.764)
  Month 6: number analyzed (Participants) | 6 | 5 | 1
  Month 6 | -6.823 (44.787) | 9.572 (24.927) | 91.640 (NA) — SD could not be calculated for a single participant.
  Month 9: number analyzed (Participants) | 8 | 3 | 1
  Month 9 | -0.019 (53.475) | 1.177 (27.654) | 89.670 (NA) — SD could not be calculated for a single participant.
  Month 12: number analyzed (Participants) | 7 | 3 | 2
  Month 12 | -40.591 (34.977) | -23.487 (30.911) | -24.905 (17.685)
  Final Study Visit (Month 49): number analyzed (Participants) | 3 | 3 | 0
  Final Study Visit (Month 49) | -28.663 (46.526) | -19.770 (74.604) |

ADVERSE EVENTS:
Time Frame: From Day 1 until the Final Study Visit (up to Month 49)
Description: TEAEs were reported for Safety population. Deaths and TEAEs were monitored together for each cohort regardless of dose administered.
Arm/Group | Zilucoplan-Cohort A (Eculizumab Naïve) | Zilucoplan-Cohort B (Eculizumab Switch) | Zilucoplan (Inadequate Responder to Eculizumab)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/6 | 2/3
Other Adverse Events (participants affected / at risk) | 9/10 | 6/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilucoplan-Cohort A (Eculizumab Naïve) (N=10) | Zilucoplan-Cohort B (Eculizumab Switch) (N=6) | Zilucoplan (Inadequate Responder to Eculizumab) (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilucoplan-Cohort A (Eculizumab Naïve) (N=10) | Zilucoplan-Cohort B (Eculizumab Switch) (N=6) | Zilucoplan (Inadequate Responder to Eculizumab) (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (7) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (9) | 2 (3) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (3) | 0 (0) | 0 (0)
Alloimmunisation (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (10) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (9) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (6) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03225287/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03225287/SAP_001.pdf